CLINICAL TRIAL: NCT05638048
Title: Effect of Precise Grip Strength Training on PICC Catheter-Related Thrombosis in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Junyan Zhao (Other)
Responsible Party: Sponsor-Investigator, Junyan Zhao, Principal investigator, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: YXLL-KY-2022(057)
Record Dates: First submitted 2022-08-24; First posted 2022-12-06 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Lung Cancer; Stomach Cancer; Breast Cancer; Liver Cancer; Colon Cancer; Rectal Cancer
Keywords: PICC；Cancer patients；Grip strength training
MeSH Terms: conditions — Lung Neoplasms; Stomach Neoplasms; Breast Neoplasms; Liver Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The control group (Active Comparator): Patients were routinely implanted with PICC and received routine health education. The content of health education included face-to-face language explanation of the whole process of catheter knowledge, issuing catheter maintenance manual, issuing ordinary grip ball and telling how to use it, and follow-up.
  Interventions: Behavioral: Health education on routine grip strength training
- Experiment 1 set (Experimental): Patients were routinely implanted with PICC, and the optimal duration-relaxation time of grip strength training was adopted on the basis of health education in the control group.
  Interventions: Behavioral: Use maximum strength grip training
- Experiment 2 set (Experimental): On the basis of control group
  1. Determine the best grip strength On the basis of the control group, color Doppler ultrasound and electronic grip force were used to record the optimal grip strength of patients to achieve effective blood flow velocity before and 24 hours after PICC insertion.
  2. Design precise grip strength training guidance program On the basis of the control group, the patients were instructed to perform grip strength training according to the determined best grip strength and the best duration of clenching and relaxation time.
  Interventions: Behavioral: Precision grip training

INTERVENTIONS:
Behavioral: Precision grip training — First determine patients for holding the ball movement should reach the effective blood flow velocity and best duration - relaxation, and USES the electronic grips and color doppler ultrasonic diagnostic apparatus, for individual patients to choose the best grip the efforts and training, to form the best grip the training plan, and observe the scheme for Peripheral central venous catheter-associated thrombosis prevention effect.
  Arms: Experiment 2 set
Behavioral: Use maximum strength grip training — Patients were routinely implanted with PICC, and on the basis of health education in the control group, the best continuous-relaxation time, frequency and maximum grip strength of patients were used for grip strength training.
  Arms: Experiment 1 set
Behavioral: Health education on routine grip strength training — Patients were routinely implanted with PICC and received routine health education. The content of health education included face-to-face language explanation of the whole process of catheter knowledge, issuing catheter maintenance manual, issuing ordinary grip ball and telling how to use it, and follow-up.
  Arms: The control group

SUMMARY:
In this study, color Doppler ultrasound diagnostic instrument and electronic grip device were used to determine the best grip strength of patients with tumor PICC catheterization, formulate precise and standardized grip strength training guidance for them, provide personalized functional exercise health education, and observe the impact of precise grip strength training guidance on Peripheral central venous catheter-associated thrombosis. To provide a reference for clinical prevention of Peripheral central venous catheter-associated thrombosis in the future.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients undergoing chemotherapy throughout their treatment in our hospital
* Patients with PICC implanted for the first time and maintained at our hospital;
* Age 18-60 years;
* Normal cognitive function;
* the clenching movement is barrier-free;
* The material and performance of PICC catheter are silicone three-way valve catheter;
* Catheter placement under the guidance of portable color Doppler ultrasound diagnostic instrument;
* Voluntarily participate and sign the informed consent form.

Exclusion Criteria:

* Patients treated with combined radiotherapy;
* Patients with coagulation dysfunction;
* Patients who need to use anticoagulant drugs due to underlying diseases;
* Puncture times more than 1 time;
* The blood flow velocity of catheterization vessel in calm state was less than 4.78cm/s.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 270 (Actual)
Dates: Start 2022-07-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Peripheral central venous catheter-associated thrombosis in patients with PICC tube | 8 weeks
  Before catheterization, 24 hours after catheterization, and weekly maintenance, color Doppler ultrasound diagnostic instrument was used to diagnose venous thrombosis (including asymptomatic thrombosis) and its classification. The patients were observed for 8 weeks.

SECONDARY OUTCOMES:
Hemodynamic changes of the patient | 8 weeks
  During weekly maintenance, color Doppler ultrasound was used to measure the blood velocity of the arm axillary vein on the side of the catheter, and the maximum blood velocity (Vmax, cm/s) was recorded.
Analysis of the influencing factors of Peripheral central venous catheter-associated thrombosis formation | 8 weeks
  By investigating the baseline data of patients, the related factors affecting the formation of PICC-CRT in patients with tumor tube in the baseline data of the same group were analyzed and compared.
Patients' satisfaction with health education after PICC catheterization | 8 weeks
  At the end of the intervention, the patients' attitude towards PICC catheterization health education questionnaire (self-made) was distributed to the study subjects, and the satisfaction of the study subjects with the health education after PICC catheterization was learned through the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Junyan Zhao, Master, Study Director — Qianfoshan Hospital; Yuanjing Qiao, Master, Principal Investigator — Shandong University of Traditional Chinese Medicine
Locations (1):
- Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided